CLINICAL TRIAL: NCT06927648
Title: CAPIVASERTIB REGULATORY POSTMARKETING SURVEILLANCE IN KOREA
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3612R00011
Record Dates: First submitted 2025-04-14; First posted 2025-04-15 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To fulfil the post-approval commitment of MFDS to conduct post-marketing surveillance, this study is designed to assess the known safety profile, identify previously unsuspected adverse reactions and to evaluate the effectiveness of Capivasertib under conditions of routine daily medical practice in Korea.

DETAILED DESCRIPTION:
The objectives of this study are to assess the safety and effectiveness of Capivasertib (hereinafter "the study drug") in a real-world practice setting for patients prescribed with the study drug under the approved local label in South Korea.

Primary Objective To assess the safety of the study drug in patients prescribed with the study drug under the approved label(s) in South Korea

Secondary Objective To assess effectiveness of the study drug in patients prescribed with the study drug under the approved label(s) in South Korea

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for and treated with the study drug according to the approved label in South Korea
* Patients who provide signed and dated written informed consent, either personally or through a legally acceptable representative.

Exclusion Criteria:

* Participation in any interventional trial during the treatment of the study drug
* Other off-label indications according to the approved label in South Korea

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently treated with or initiating the study drug under approved local label and conditions of routine daily medical practice in South Korea will be included in the study. This study will be conducted using a total surveillance method to investigate the safety and effectiveness of all patients being treated with the study drug.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs)·Adverse Drug Reactions (ADRs) Serious Adverse Events (SAEs)·Adverse Drug Reactions (SADRs) Unexpected Adverse Events (AEs)·Adverse Drug Reactions (ADRs) | For about 12 months from the first dose of the study drug unless they withdraw consent, are lost to follow-up, experience disease progression, or die. 30 days addtional follow up in case of not completing 12 months.
  The safety assessment should include all undesirable changes in medical findings (including clinical test findings) noted during medical visits as required by local practice guidelines, as well as all AEs associated with the study drug administration.

SECONDARY OUTCOMES:
Real-world progression free survival (rwPFS) | For about 12 months from the first dose of the study drug unless they withdraw consent, are lost to follow-up, experience disease progression, or die
  Real-world progression free survival (rwPFS) for patients will be evaluated by routine clinical practice of the investigators. rwPFS will be defined as the time from first dose of the study drug until the date of disease progression or death (by any cause in the absence of progression) regardless of whether the subject withdraws from therapy or receives another anti-cancer therapy prior to progression.Subjects who have not progressed or died at the time of analysis will be censored at the date of their last follow-up assessment.

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Research Site, Busan
  - Research Site, Daejeon
  - Research Site, Goyang-si
  - Research Site, Guri-si
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/